CLINICAL TRIAL: NCT00235248
Title: Prevention of New Vascular Events in Patients With Brain Infarction or Peripheral Embolism and Thoracic Aortic Plaques ≥ 4 mm in Thickness in the Aortic Arch or Descending Aortic Upstream to the Embolized Artery
Brief Title: Aortic Arch Related Cerebral Hazard Trial (ARCH)
Acronym: ARCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P991205
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Brain Infarction; Transient Ischemic Attack; Embolism
Keywords: TIA/Brain infarct; and plaque>4mm in the aortic arch; Or peripheral embolism; and plaque>4 mm in the thoracic aorta
MeSH Terms: conditions — Brain Infarction; Ischemic Attack, Transient; Embolism | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel-aspirin (Experimental): Clopidogrel-aspirin
  Interventions: Drug: Clopidogrel-aspirin
- Warfarin (Active Comparator): Warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Warfarin
  Arms: Warfarin
Drug: Clopidogrel-aspirin — Clopidogrel-aspirin
  Arms: Clopidogrel-aspirin

SUMMARY:
The ARCH is a controlled trial with a sequential design and with a prospective, randomized, open-label, blinded-endpoint (PROBE) methodology. The objective is to compare the efficacy and tolerance (net benefit) of two antithrombotic strategies in patients with atherothrombosis of the aortic arch and a recent (less than 6 months) cerebral or peripheral embolic event.

Hypothesis:

The association of clopidogrel 75 mg/d plus aspirin 75 mg/d is 25% more effective than an oral anticoagulant (target International Normalized Ratio [INR] 2 to 3) in preventing brain infarction, brain hemorrhage, myocardial infarction, peripheral embolism, and vascular death.

DETAILED DESCRIPTION:
Patients with Transient Ischemic attack or brain infarction of unknown cause (no ipsilateral internal carotid artery origin stenosis greater than 70%, no ipsilateral severe intracranial stenosis of an artery supplying the infarcted area, no definite cardiac source of embolism) in the preceding 6 months and atherosclerotic plaques.

≥ 4 mm in the aortic arch, or patients with a peripheral event (e.g. renal infarct) in the preceding 6 months and plaque ≥ 4 mm in the thoracic aorta above the origin of the embolized artery.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes aged ≥ 18 years with the following 4 inclusion criteria:

* One of the 3 following ischemic events in the preceding 6 months:

  * Transient ischemic attack (TIA)
  * Non-disabling brain infarcts:

    * Inclusion within 6 months after onset
    * Duration of symptoms and signs greater than 24 hours
    * Neurological signs at the time of randomization with a Rankin Scale grade 3 or less
    * With normal computed tomography (CT) scan or CT scan showing a brain infarct (even hemorrhagic infarct)
  * Peripheral embolism
* Atherosclerotic plaque in the thoracic aorta is defined as wall thickness ≥ 4 mm where the protruding material is the largest, measured at transesophageal echocardiography with multiplane transducer or a plaque less than 4 mm but with mobile component.
* Informed consent signed
* Life expectancy > 3 years

Exclusion Criteria:

* Other causes of embolism:

  * Cardiac: endocarditis, atrial fibrillation, intra-cardiac thrombus, valvular prosthesis, rheumatic valvulopathy, left ventricular aneurysm, or ejection fraction less than 25%
  * Atherosclerotic stenosis ipsilateral to the embolic territory: internal carotid artery stenosis greater than 70%, or severe (judgment of the investigator) intracranial stenosis, or scheduled carotid endarterectomy (in that case inclusion is possible 30 days after the procedure)
  * Uncommon causes: dissection, vasculitis, procoagulant state, or sickle cell disease
* Other exclusion criteria:

  * Intercurrent illness with life expectancy less than 36 months
  * Pregnancy and non-menopausal women
  * Unwillingness to participate
  * Poor medication compliance expected
  * Toxicomania
  * Absolute indication for anticoagulant therapy (e.g. atrial fibrillation, intracardiac thrombus, prosthetic valve)
  * Scheduled for carotid endarterectomy (randomization is possible 30 days after endarterectomy)
* CT scan with an intracranial lesion other than brain infarction (space occupying mass, intracranial hemorrhage)
* Transesophageal echocardiography (TEE) with plaque ≥ 4 mm in thickness distal to the supposed embolized artery (judgement of the investigator).
* Contraindication to clopidogrel, aspirin, and oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2002-02; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
New vascular events assessed every 4 months including stroke, myocardial infarction (MI), peripheral events, and vascular death | every 4 months
  New vascular events assessed every 4 months including stroke, myocardial infarction (MI), peripheral events, and vascular death

SECONDARY OUTCOMES:
Recurrent brain infarction | during the trial
  Recurrent brain infarction
brain infarction and transient ischemic attack (TIA) | during the studing
  brain infarction and transient ischemic attack (TIA)
new vascular events and revascularization procedure | during the trial
  new vascular events and revascularization procedure
vascular death | during the trial
  vascular death
death from all causes | during the trial
  death from all causes
combination of primary end-point and TIA | during the trial
  combination of primary end-point and TIA
revascularization procedures | during the trial
  revascularization procedures
urgent rehospitalization for ischemic | during the trial
  urgent rehospitalization for ischemic

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Amarenco, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- National Stroke Research Institute-Austin Health, Heidelberg Heights, Australia
- Bichat Hospital Head of Neurology Department, Paris, France

REFERENCES:
- [Derived] Amarenco P, Davis S, Jones EF, Cohen AA, Heiss WD, Kaste M, Laouenan C, Young D, Macleod M, Donnan GA; Aortic Arch Related Cerebral Hazard Trial Investigators. Clopidogrel plus aspirin versus warfarin in patients with stroke and aortic arch plaques. Stroke. 2014 May;45(5):1248-57. doi: 10.1161/STROKEAHA.113.004251. Epub 2014 Apr 3. PMID 24699050